CLINICAL TRIAL: NCT04883450
Title: PRedictiOn Algorithms for the DeTECTion of Early Stage Pancreatic Cancer
Acronym: PRO-TECT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kaiser Permanente (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 12135; R01CA230442 (NIH)
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma (PDAC)
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood (plasma, serum and Buffy coat) and Urine samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Risk of pancreatic cancer: Subjects with an increased predicted 18-month risk of pancreatic cancer
  Interventions: Diagnostic Test: Magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging (MRI) — All enrolled participants will undergo magnetic resonance imaging (MRI) at their Baseline and 18-Month follow-up visit

SUMMARY:
Conduct a prospective study to assess the accuracy of a pancreatic cancer risk prediction model.

DETAILED DESCRIPTION:
The goal of this study is to establish a platform for development and implementation of a data-driven risk model for detection of early stage pancreatic cancer within an integrated health care setting. Patients at increased risk for pancreatic cancer as identified by the risk model will be invited to participate in a prospective study to assess the accuracy of this approach for detection of early stage pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have 6 months of membership
2. Patient has a measure for weight, Hemoglobin A1C, and Alanine transaminase (ALT) within the past 6 months
3. Patient must have an increased predicted 18-month risk of pancreatic cancer based on the PRO-TECT model
4. Speaks English or Spanish

Exclusion Criteria:

1. Previous or current history of pancreatic cancer
2. Metastatic cancer
3. Current active cancer or undergoing chemotherapy for cancer
4. Currently pregnant or breastfeeding
5. Class IV heart failure
6. Cirrhosis with ascites and/or varices
7. Currently in a skilled nursing facility or under hospice care
8. Has metal parts or implanted devices in the body, such as a pacemaker, defibrillator, or shrapnel
9. End stage renal disease
10. Cognitive impairment such that the person is unable to provide informed consent

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kaiser Permanente Southern California with at least 12 months prior to recruitment
Sampling Method: Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of pancreatic ductal adenocarcinoma (PDAC) in the high predicted risk group | 18-Month
  Enrolled subjects will be followed for 18 months to determine the incidence rate of PDAC

CONTACTS AND LOCATIONS:
Overall Officials: Bechien U Wu, MD, MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Southern California, Pasadena, California, United States

IPD SHARING:
Plan to Share IPD: No